CLINICAL TRIAL: NCT02536534
Title: (e-MOTION PH) Electronic - Activity Level Monitoring Pilot in Pulmonary Hypertension
Brief Title: Electronic Activity Level Monitoring Pilot in Pulmonary Hypertension
Acronym: e-MOTION PH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17926; DBOX 2014/00466 (Other: Company internal)
Record Dates: First submitted 2015-08-10; First posted 2015-09-01 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension (PAH); Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with PAH and CTEPH: Patients diagnosed with symptomatic Pulmonary Arterial Hypertension (PAH) or Chronic Thromboembolic Pulmonary Hypertension (CTEPH) and stable on optimal medical therapy who meet the study's eligibility criteria
  Interventions: Other: Correlation assessment

INTERVENTIONS:
Other: Correlation assessment

SUMMARY:
Evaluate the correlation between activity level (monitored by Fitbit Flex remote activity tracker) and 6-minute walk distance (6MWD) (performed by investigator) in patients with Pulmonary Arterial Hypertension (PAH) or Chronic Thromboembolic Pulmonary Hypertension (CTEPH) over 6 months in routine clinical practice settings.

DETAILED DESCRIPTION:
Remote patient monitoring can lead to improved patient outcomes, including improved quality of life, reduced readmissions, earlier treatment for symptoms detected prior to schedule in-office follow-up visits, improved communications with care providers, increased participation in self-management of disease, and an improved knowledge of their medical conditions . In patients with PAH, daily activity level, as measured using a physical activity monitor for seven consecutive days, correlated with 6-minute walk distance (6MWD). The monitor used in the aforementioned PAH study was positioned on the patients' right upper arm with an armband, as opposed to the more popular and more comfortable wristbands used today, such as the Fitbit Flex. Although the aforementioned PAH study did show a correlation between activity level monitoring and 6MWD, the patients were monitored for only seven days. It is still unknown whether this correlation would exist over a longer trial period and whether patients, their caregivers, and clinicians would find activity level monitoring useful in helping manage PH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a diagnosis of Pulmonary Arterial Hypertension (PAH); or inoperable, persistent or recurrent Chronic Thromboembolic Pulmonary Hypertension (CTEPH),
* Age ≥ 18 years,
* Baseline 6 Minute Walk Distance (6MWD) a minimum of 250 meters or maximum 450 meters, (ensure significant Pulmonary Hypertension(PH) without limiting their participation in the trial)
* WHO Functional Class II or III,
* Clinically stable patient defined as within the last 12 months (minimum of 3 months) prior to enrollment, there was no:

  * decline in World Health Organization (WHO) Function class or,
  * decline in 6MWD by 15% or,
  * change of oral PAH/CTEPH therapy (may have flexible diuretics/anticoagulation) or,
  * Introduction of parenteral Prostacyclin Analog (PCA) treatment.
* Patients provide written informed consent, are able to understand and follow instructions.

Exclusion Criteria:

* Hypersensitivity to nickel (present in the clasp of the FitBit Flex's band),
* Medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator,
* Enrolled in pulmonary rehabilitation program within last 6 months,
* Participating in an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian patients are eligible for the study if they have been diagnosed with symptomatic Pulmonary Arterial Hypertension (PAH) or Chronic Thromboembolic Pulmonary Hypertension (CTEPH) and are stable on optimal medical therapy and who meet the study's eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) | At baseline
  (performed by investigator)
6-minute walk distance (6MWD) | At 3 months
  (performed by investigator)
6-minute walk distance (6MWD) | At 6 months
  (performed by investigator)
Number of steps per day | At baseline
  (monitored by Fitbit Flex)
Number of steps per day | At 3 months
  (monitored by Fitbit Flex)
Number of steps per day | At 6 months
  (monitored by Fitbit Flex)

SECONDARY OUTCOMES:
Change in quality of life recorded by patient questionnaire Living with Pulmonary hypertension Questionnaire (LPH) | At baseline, 3 months and 6 months
Change in compliance with medication using the Moriky´s Questionnaire | At baseline, 3 months and 6 months
Change in World Health Organization (WHO) functional Class recorded by investigator in conjunction with the 6MWD | At baseline, 3 months and 6 months
Change in Borg Dyspnea value recorded by investigator in conjunction with the 6MWD | At baseline, 3 months and 6 months
Healthcare provider Satisfaction and Usability questionnaire | At 3 months and 6 months
Caregiver Satisfaction and Usability questionnaire | At 3 months and 6 months
Patient Satisfaction and Usability questionnaire | At 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Canada